CLINICAL TRIAL: NCT04787198
Title: Investigating Composite Biomarkers for Pain Catastrophizing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Laura Petrini, Associate Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20200095
Record Dates: First submitted 2021-02-16; First posted 2021-03-08 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypertonic saline (Experimental)
  Interventions: Drug: hypertonic saline
- isotonic saline (Placebo Comparator)
  Interventions: Drug: isotonic saline

INTERVENTIONS:
Drug: hypertonic saline — The site of injections will be determined by palpation of the contracted First Dorsal Interosseus (FDI) muscle. The skin will be cleaned with alcohol before injection. A bolus injection of hypertonic saline (7% NaCl) will be administered to the FDI muscle using a 1 mL syringe with a disposable needle (27G), and 30 the volume of the bolus will be 0.2 mL .
  Arms: hypertonic saline
Drug: isotonic saline — The site of injections will be determined by palpation of the contracted First Dorsal Interosseus (FDI) muscle. The skin will be cleaned with alcohol before injection. A bolus injection of 0.2 mL isotonic saline (9 mg/mL) will be administered to the FDI muscle as control.
  Arms: isotonic saline

SUMMARY:
Pain is a complex, multidimensional, and subjective experience; and although, investigators use a single word "pain", to describe our perception, multiple mechanisms contribute to the generation and maintenance of pain. To help diagnosing and improving pain management, there is a need for developing tools. These tools may include measurements of substances, or biomarkers, in the blood; e.g. small molecules called microRNA and proteins. In these experiments, the investigators would like to investigate how the psychological response to stress and pain alters the impulses in the brain and the content of microRNA and proteins in the blood. The future aim is to identify patients in high risk of developing and maintaining chronic pain and to be able to treat chronic pain efficiently.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women in the age 18-80 years
* Speak and understand English

Exclusion Criteria:

* Acute and chronic pain
* Pregnancy or breastfeeding
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Present or previous history of neurological, dermatological, immunological, musculoskeletal, cardiac disorder or mental illnesses that may affect the results (e.g. Neuropathy, muscular pain in the upper extremities, etc.)
* Focal and generalized seizure
* Surgery or any other therapy for epilepsy
* Present or previous AEDs (anti-epileptic drugs) administration
* Present or previous use of epileptic devices (<1 year prior the enrolment)
* Lack of ability to cooperate
* Current use of medications that may affect the trial, such as antipsychotics and pain killers as well as systemic or topical steroids and anti-inflammatory drugs.
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Oscillations of the main electroencephalogram (EEG) frequency | 10 minutes of recording before isotonic/hypertonic injection
  Electroencephalographic (EEG) recording will be performed placing a 64-electrodes cap over the scalp according to the 10-20 international system. Oscillations of the main EEG frequency bands (delta, alpha, beta, gamma) from the frontal and parietal lobes will be detected and correlated to the individual pain rate as well as the dimensions of the psychological questionnaires.
Oscillations of the main electroencephalogram (EEG) frequency | 10 minutes of recording after isotonic/hypertonic injection
  Electroencephalographic (EEG) recording will be performed placing a 64-electrodes cap over the scalp according to the 10-20 international system. Oscillations of the main EEG frequency bands (delta, alpha, beta, gamma) from the frontal and parietal lobes will be detected and correlated to the individual pain rate as well as the dimensions of the psychological questionnaires.
Perturbation of the electroencephalogram (EEG) rhythms | 10 minutes of recording before isotonic/hypertonic injection
  Electroencephalographic (EEG) recording will be performed placing a 64-electrodes cap over the scalp according to the 10-20 international system. Perturbation of the above-mentioned EEG rhythms will be measured in response to the hypertonic/isotonic saline injection and compared to a resting state baseline recording.
Perturbation of the electroencephalogram (EEG) rhythms | 10 minutes of recording after isotonic/hypertonic injection
  Electroencephalographic (EEG) recording will be performed placing a 64-electrodes cap over the scalp according to the 10-20 international system. Perturbation of the above-mentioned EEG rhythms will be measured in response to the hypertonic/isotonic saline injection and compared to a resting state baseline recording.
Collection of blood samples | time 0 (baseline)
  Whole blood samples (5 mL per each time point, a total of 20 mL per subject) will be collected into SST™ II Advance Serum Separation Tubes containing anticoagulant EDTA.
Collection of blood samples | Time 1 (3 hours)
  Whole blood samples (5 mL per each time point, a total of 20 mL per subject) will be collected into SST™ II Advance Serum Separation Tubes containing anticoagulant EDTA.
Collection of blood samples | time 2 (24 hours)
  Whole blood samples (5 mL per each time point, a total of 20 mL per subject) will be collected into SST™ II Advance Serum Separation Tubes containing anticoagulant EDTA.
Collection of blood samples | time 3 (48 hours)
  Whole blood samples (5 mL per each time point, a total of 20 mL per subject) will be collected into SST™ II Advance Serum Separation Tubes containing anticoagulant EDTA.
Collection of blood samples | time 4 (72 hours)
  Whole blood samples (5 mL per each time point, a total of 20 mL per subject) will be collected into SST™ II Advance Serum Separation Tubes containing anticoagulant EDTA.
MicroRNAs (miRNAs) expression analysis | time 0 (baseline)
  From the blood samples previously collected, miRNA will be isolated for a subsequent miRNA library preparation. Subsequently, extracted miRNA will be reversely transcribed, and cDNA will be used for total miRNAs sequencing.
MicroRNAs (miRNAs) expression analysis | time 1 (3 hours)
  From the blood samples previously collected, miRNA will be isolated for a subsequent miRNA library preparation. Subsequently, extracted miRNA will be reversely transcribed, and cDNA will be used for total miRNAs sequencing.
MicroRNAs (miRNAs) expression analysis | time 2 (24 hours)
  From the blood samples previously collected, miRNA will be isolated for a subsequent miRNA library preparation. Subsequently, extracted miRNA will be reversely transcribed, and cDNA will be used for total miRNAs sequencing.
MicroRNAs (miRNAs) expression analysis | time 3 (48 hours)
  From the blood samples previously collected, miRNA will be isolated for a subsequent miRNA library preparation. Subsequently, extracted miRNA will be reversely transcribed, and cDNA will be used for total miRNAs sequencing.
MicroRNAs (miRNAs) expression analysis | time 4 (72 hours)
  From the blood samples previously collected, miRNA will be isolated for a subsequent miRNA library preparation. Subsequently, extracted miRNA will be reversely transcribed, and cDNA will be used for total miRNAs sequencing.
Proteome analysis | time 0 (baseline)
  From the blood samples previously collected, the protein concentration will be determined. Protein sequencing will be done using mass spectrometers.
Proteome analysis | time 1(3 hours)
  From the blood samples previously collected, the protein concentration will be determined. Protein sequencing will be done using mass spectrometers.
Proteome analysis | time 2 (24 hours)
  From the blood samples previously collected, the protein concentration will be determined. Protein sequencing will be done using mass spectrometers.
Proteome analysis | time 3 (48 hours)
  From the blood samples previously collected, the protein concentration will be determined. Protein sequencing will be done using mass spectrometers.
Proteome analysis | time 4 (72 hours)
  From the blood samples previously collected, the protein concentration will be determined. Protein sequencing will be done using mass spectrometers.
Metabolome analysis | time 0 (baseline)
  From the blood samples previously collected. Metabolites will be investigated and identified by a 4D feature finding using Metaboscape.
Metabolome analysis | time 1(3 hours)
  From the blood samples previously collected. Metabolites will be investigated and identified by a 4D feature finding using Metaboscape.
Metabolome analysis | time 2 (24 hours)
  From the blood samples previously collected. Metabolites will be investigated and identified by a 4D feature finding using Metaboscape.
Metabolome analysis | time 3 (48 hours)
  From the blood samples previously collected. Metabolites will be investigated and identified by a 4D feature finding using Metaboscape.
Metabolome analysis | time 4 (72 hours)
  From the blood samples previously collected. Metabolites will be investigated and identified by a 4D feature finding using Metaboscape.
Plasma cortisol levels measurement | time 0 (baseline)
  From the blood samples previously collected, plasma levels of cortisol will be evaluated through enzyme-linked immunosorbent assay (ELISA).
Plasma cortisol levels measurements | time 1(3 hours)
  From the blood samples previously collected, plasma levels of cortisol will be evaluated through enzyme-linked immunosorbent assay (ELISA).
Plasma cortisol levels measurements | time 2 (24 hours)
  From the blood samples previously collected, plasma levels of cortisol will be evaluated through enzyme-linked immunosorbent assay (ELISA).
Plasma cortisol levels measurements | time 3 (48 hours)
  From the blood samples previously collected, plasma levels of cortisol will be evaluated through enzyme-linked immunosorbent assay (ELISA).
Plasma cortisol levels measurements | time 4 (72 hours)
  From the blood samples previously collected, plasma levels of cortisol will be evaluated through enzyme-linked immunosorbent assay (ELISA).
Plasma Interleukin-6 (IL-6) levels measurements | time 0 (baseline)
  From the blood samples previously collected, plasma levels of IL-6 will be evaluated through enzyme-linked immunosorbent assay (ELISA).
Plasma Interleukin-6 levels measurements | time 1(3 hours)
  From the blood samples previously collected, plasma levels of IL-6 will be evaluated through enzyme-linked immunosorbent assay (ELISA).
Plasma Interleukin-6 levels measurements | time 2 (24 hours)
  From the blood samples previously collected, plasma levels of IL-6 will be evaluated through enzyme-linked immunosorbent assay (ELISA).
Plasma Interleukin-6 levels measurements | time 3 (48 hours)
  From the blood samples previously collected, plasma levels of IL-6 will be evaluated through enzyme-linked immunosorbent assay (ELISA).
Plasma Interleukin-6 levels measurements | time 4 (72 hours)
  From the blood samples previously collected, plasma levels of IL-6 will be evaluated through enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Measuring Pain using VAS | 20 minutes
  The subject will rate the pain intensity continuously for 20 minutes and VAS will start from zero (0), representing no pain, and will end at one hundred (100) representing worst pain imaginable.

OTHER OUTCOMES:
Pain Catastrophizing Scale (PCS) questionnaire | time 0 (baseline)
  The PCS assesses negative and exaggerated coping concerning anticipated or experienced painful stimuli. Thirteen items have to be answered on a 5-points Likert-type scale from 0 (non at all) to 4 (all the time).
Positive and Negative Affect Schedule (PANAS) questionnaire | time 0 (baseline)
  The PANAS measures positive affects (PA) dimensions ( "the extent to which a person feels active, enthusiastic, and alert") and negative affects (NA) dimensions (a condition of "general distress and unpleasable engagement"). Twenty words are associated with the subject's current feelings and have to be rated on a 5-points Likert-type scale from 1 (non at all) to 5 (extremely).
Reinforcement Sensitivity Theory - Personality Questionnaire (RST-PQ). | time 0 (baseline)
  The RST-PQ contains the following subscales:
  * Fight-Flight-Freeze System (FFFS, 10 items), related to active avoidance of adverse stimuli;
  * Behavioral Inhibition System (BIS, 23 items), related to anxiety and passive avoidance of adverse stimuli;
  * Behavioral Approach System (BAS, 32 items), it reflects reward interest, reward reactivity, impulsivity.
  In total, 65 items have to be answered on a 4-points Likert-type scale, from 1 (non at all) to 4 (highly).
State-Trait Anxiety Inventory - Form Y (STAI-Y) | time 0 (baseline)
  The STAI-Y questionnaire measures two types of anxiety, the state and the trait anxiety, as well as the severity of the overall anxiety level. The questionnaire is divided into two sections of 20 items each to be rated on a 4-points Likert-type scale from 1 (non at all) to 4 (very much).
Heart rate assessment | time 0 (baseline)
  An electrocardiogram (ECG) will be recorded with a standard 3-lead montage (one electrode on each wrist and the third on the left ankle)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Petrini, PhD, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No